CLINICAL TRIAL: NCT03147755
Title: Prevalence, Risk Factors and Complications of Oropharyngeal Dysphagia in Stroke Patients
Acronym: Marato-11
Status: Completed | Type: Observational
Sponsor: Pere Clave (Other)
Responsible Party: Sponsor-Investigator, Pere Clave, MD, PhD, Hospital de Mataró
Organization: Hospital de Mataró (Other)
Other Study IDs: 17/11
Record Dates: First submitted 2017-05-04; First posted 2017-05-10 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Deglutition Disorders
Keywords: stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dysphagia: Patients with stroke associated dysphagia
  Interventions: Other: No intervention
- No dysphagia: Patients without stroke associated dysphagia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Oropharyngeal dysphagia (OD) is a common morbidity after stroke that disrupts swallowing physiology. The investigators aimed at evaluating the prevalence of oropharyngeal dysphagia (OD) after stroke and analysing the risk factors and associated complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to hospital with confirmed stroke diagnosis; signed informed consent

Exclusion Criteria:

* previous diagnosis of OD; transient ischemic attack; and being transferred from another hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with clinical suspicion of stroke
Sampling Method: Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year
  OD mortality rates has been assessed

IPD SHARING:
Plan to Share IPD: No